CLINICAL TRIAL: NCT03566121
Title: Prediction of the Severity of Female SUI by Measuring New Static and Dynamic Ultrasound Parameters of the Urethra
Acronym: PRESIUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018/01
Record Dates: First submitted 2018-06-12; First posted 2018-06-21 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Incontinence, Urinary
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continent women (Other): Women with ICI-Q=0 Pelvic ultrasound / Urodynamic ultrasound
  Interventions: Other: Pelvic ultrasound / Urodynamic ultrasound
- Incontinent women (Experimental): Women with ICI-Q≥1 Pelvic ultrasound / Urodynamic ultrasound
  Interventions: Other: Pelvic ultrasound / Urodynamic ultrasound

INTERVENTIONS:
Other: Pelvic ultrasound / Urodynamic ultrasound — Gynecological consultation: calculating the score ICI-Q Ultrasound consultation: pelvic ultrasound Urodynamic ultrasound during a Valsalva manoeuvers

SUMMARY:
This study aims to evaluate the correlation of the ultrasonic functional length of the urethra and the incontinence urinary disorder (IUD). The goal is to predict the severity of the IU by measuring new static and dynamic ultrasound parameters of the urethra.

DETAILED DESCRIPTION:
The urinary incontinence is a disorder which affects 25 to 45% of women. Nowadays, the role of urethral tissue in IUD is not explored although well viewed in perineal ultrasound. Our actual knowledge demonstrates that urodynamic ultrasound is reliable to establish the bladder neck mobility. And the posterior urethral wall mobility was often associated to the stress urinary incontinence. Two elements appeared to indicate the elasticity of the urethral environment: functional length urethral variation and urethral closure angle variation during Valsalva manoeuvres compared to rest. This study aims to evaluate the correlation of the ultrasonic functional length of the urethra and the incontinence urinary disorder for the purpose to predict the severity of this syndrome.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged over 18 years addressed to pelvic ultrasound

Exclusion Criteria:

* Pregnant
* Post-partum (under 6 month of childbirth)
* Operated for a genitourinary prolapse or/and urinary incontinence
* Utero vaginal symptomatic prolapse
* Overactive bladder ± UI by
* Dysuria
* Severe deep pelvic endometriosis
* Respiratory failure (Unable to perform the Valsalva manoeuvres)
* History of pelvic cancer
* Unable to understand the information communicated

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-07-13 (Actual)

PRIMARY OUTCOMES:
Measurement of ultrasonic urethral length | From 3 to 11 days after gynecological consultation
  LT total length LF functional length LE funnel urethral length Measurement of the angle between proximal and distal urethra

CONTACTS AND LOCATIONS:
Overall Officials: Georges BADER, MD, Principal Investigator — CMC Hartmann
Locations (2):
- France (2):
  - CMC Hartmann, Neuilly-sur-Seine
  - Centre Echographie Obstétricale, Paris

IPD SHARING:
Plan to Share IPD: No